CLINICAL TRIAL: NCT00220038
Title: Genetic Basis of Specific Anosmias
Brief Title: Experiments to Test How and Why the Sense of Smell Differs Between People
Status: Completed | Type: Observational
Sponsor: Rockefeller University (Other)
Responsible Party: Sponsor
Other Study IDs: LVO-0539
Record Dates: First submitted 2005-09-21; First posted 2005-09-22 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2012-01

CONDITIONS: Specific Anosmias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Normal: 700 healthy adult volunteers will be drawn from the New York City area
  Interventions: Behavioral: smell tests

INTERVENTIONS:
Behavioral: smell tests — subjects are instructed to sniff two vials, one containing the solvent, the other a dilution of the odorant. They are asked to scan the vial with the stronger odor.

SUMMARY:
The ability to smell varies greatly between different individuals. Some people are unable to detect an odor that most people can smell. It is not known what causes these individual differences. Humans have about 1000 genes for odorant receptors that bind and detect odor molecules. It has been shown that some of these genes exist in two forms: a functional one and one that has been mutated and is therefore no longer functional. We think that people who can not smell a specific odor may carry the non-functional form of the gene for the receptor that detects the odor molecule. To test this hypothesis we want to find people who can not detect a specific smell and then compare their odorant receptor genes with those of people who can smell the odor.

DETAILED DESCRIPTION:
The enjoyment of a fine wine, the odor of a ripe cheese, the memory of a long-lost grandmother brought back by the scent of her perfume, or the alarm we feel when we smell smoke are all produced by a functioning olfactory system. Interestingly, there are enormous individual differences in how we interpret these smells. Given almost any odor, some people will find it pleasant, others unpleasant. Ripe cheese or garlic may smell delicious to some, but repulsive to others. The scientific basis of this variation has not been well-studied. Despite the clear evidence for culture-based preferences for food and aromas, the nature-versus-nurture debate for smell remains unresolved. We believe there may be a genetic basis for our unique senses of smell. For example, some of us can smell methanethiol, the metabolite that is excreted in our urine after eating asparagus, whereas other people cannot. The Rockefeller University Smell Study seeks to recruit 400 normal subjects to track down the genetic basis of how we perceive smells. The study consists of up to two visits, each lasting up to 4 hours, in which we will test your perception of a variety of smells. On your first visit there will be a small blood sample taken (8.5 millileters) and your height and weight will be measured. If you are a woman of child-bearing age, we will ask you to provide a urine sample to test for pregnancy. If you are pregnant, you will not be permitted to participate in our study. You will fill out a short survey that asks some questions about yourself, your household, your personal habits, and your sense of smell. You will perform three different types of smell tests. In the first, you will be given two vials at a time and asked to tell us which contains an odor. In the second type of test, you will be asked to describe carefully your impression of three different odors. In the third type of test, you will be asked to rate odors according to their strength and pleasantness. All odorants will be presented to you in glass jars. You will be asked to smell odors in several hundred jars.

ELIGIBILITY:
Inclusion Criteria:

18 years or older,

Male and Female

Normal sense of smell

-

Exclusion Criteria:

Not pregnant

No history of nasal illness or surgery

No seasonal allergies-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 700 healthy normal volunteers will be recruited from the New York City area
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2004-05; Primary Completion 2007-01 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie B. Vosshall, PHD, Principal Investigator — Rockefeller University
Locations (1):
- Rockefeller University Hospital, New York, New York, United States